CLINICAL TRIAL: NCT04855825
Title: Investigating the Effects of Wearable Robotic Exoskeleton for Improving Mobility and Cognition in Persons With MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, Ghaith J. Androwis, Ph.D., Assistant Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-983-17
Record Dates: First submitted 2018-06-18; First posted 2021-04-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic; Motility Disorder; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic Exoskeleton Therapy (Experimental): Gait rehabilitation provided using a wearable robotic exoskeleton
  Interventions: Device: Robotic Exoskeleton Rehabilitation
- Conventional Gait Therapy (Active Comparator): Gait rehabilitation provided using traditional gait therapy under the supervision of a licensed PT
  Interventions: Other: Conventional Gait Therapy

INTERVENTIONS:
Device: Robotic Exoskeleton Rehabilitation — Participants will be randomly assigned to one of the two groups. Each participant will receive 8 sessions of gait rehabilitation and therapy via traditional therapy techniques of using the robotic exoskeleton. This training will be provided by a licensed physical therapist.
  Arms: Robotic Exoskeleton Therapy
Other: Conventional Gait Therapy — Participants will be randomly assigned to one of the two groups. Each participant will receive 8 sessions of gait rehabilitation and therapy via traditional therapy techniques of using the robotic exoskeleton. This training will be provided by a licensed physical therapist.
  Arms: Conventional Gait Therapy

SUMMARY:
The purpose of this research study is to evaluate the usefulness of a wearable robotic exoskeleton device (Ekso-GT), to improve learning and memory, and gait therapy in persons with walking disability due to Multiple Sclerosis. The study will evaluate the mobility, learning and memory, and walking abilities of individuals with multiple sclerosis who went through the traditional as compared to others who used the robotic exoskeleton as part of their therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with multiple sclerosis.
* Be determined by the study staff to have moderate to severe difficulty walking but still be able to walk while using the robotic exoskeleton.
* Have some difficulty thinking and problem solving as determined by my performance on a special test that I will take during the screening visit.
* Be between the ages of 18 and 75.
* Be free from flair ups of my MS Symptoms for at least one month prior to testing.
* Discuss with study staff how to maintain a constant level of my spasticity medication (for example baclofen) throughout the study.
* Be able to walk (with the use of one or more assistive device if needed).
* Have English as my primary language.
* Be able to physically fit into the exoskeleton device: height between 60 and 76", weight under 220 lbs.
* Be able to tolerate upright standing for 30 minutes with assistance if needed.
* Have normal joint range of motion for walking as determined by study staff.
* Have sufficient strength to use the hemiwalker, bilateral canes or walker while wearing the RE.
* Have stable blood pressure.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures and follow directions and commands, verbal instructions, and follow-up requirements.

Exclusion Criteria:

* Have a history of head injury, stroke, seizures, or any other significant neurological history other than MS.
* Have a high degree of difficulty in thinking and problem solving that prevents me from participating in the study as determined by my performance on a special test taken during the screening visit.
* Be currently taking steroids, benzodiazepines, antipsychotics, and/or neuroleptics as determined by study staff review of my medications.
* Be pregnant.
* Be completely reliant on a wheelchair.
* Have joint contracture or spasticity of any limb that limits normal range of motion during walking with assistive devices as determined by study staff.
* Have skin issues that would prevent wearing the RE.
* Have pressure sore stage 2 or higher located in an area that would negatively affect weight bearing, harness fit, or therapist assistance.
* Have orthopedic issues or history that will interfere with walking or limit the range of motion of the lower limbs (e.g., knee replacement, inflammation)
* Have been hospitalized for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Have any other medical conditions that my doctor or physical therapist feels would affect my ability to use the robotic device.
* Have a pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* Have dental implants- I should discuss any dental implants with the investigators.
* Have been told by my doctor that it is unsafe for me to have a regular MRI as part of my medical care.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Distance walked in a specific time duration | approximately 12 weeks
  The distance walked (meters) in 6 minutes is measured. This is following the 6-minute walk test (6MWT) procedure to measure walking endurance. The 6MWT is is a valid and reliable test of endurance walking performance in persons with MS.
  Participants are instructed to walk as fast and as far as possible for 6 minutes within a single corridor and performing 180° turns.
Neuropsychological measures of thinking | approximately 12 weeks
  Processing speed and cognition outcomes, including: The Symbol Digit Modalities Test (SDMT) represents the primary CPS outcome in the current proposal. This test involves the conversion of a set of simple geometric designs into an oral response. It has been demonstrated to be sensitive to the presence of brain damage in numerous studies. The SDMT requires the examinee to substitute a number for a randomized presentation of a geometric figure. The appropriate number is shown in a key containing the Arabic numbers 1 through 9, each paired with a different geometric figure. The total number of correct responses in 90 seconds is the primary outcome of the SDMT.
Brain scans | approximately 12 weeks
  Participants will undergo neuroimaging scans of the brain to acquire structural imaging of the brain using Magnetic resonance imaging (MRI).
  The MRI instrument that will be used is an FDA-approved Siemens Skyra 3T clinical imager housed in the Rocco Ortenzio Neuroimaging Center at Kessler Foundation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided